CLINICAL TRIAL: NCT05308602
Title: A Randomized, Double-blinded, Active-controlled Phase II Clinical Study to Evaluate the Immunogenicity and Safety of SCTV01C (A Bivalent SARS-CoV-2 Trimeric Spike Protein Vaccine) and SCTV01E (A COVID-19 Alpha/Beta/Delta/Omicron Variants S-Trimer Vaccine) in Population Aged ≥12 Years and Previously Unvaccinated
Brief Title: A Study to Evaluate the Immunogenicity and Safety of SCTV01C and SCTV01E (Two Recombinant Protein COVID-19 Vaccines) in Population Aged ≥12 Years
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: There was not a need any more.
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SCTV01C/E-02-In-Laos-1
Record Dates: First submitted 2022-02-15; First posted 2022-04-04 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2022-03

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: COVID-19; SARS-CoV-2 infection; Vaccine
MeSH Terms: conditions — COVID-19 | interventions — SCTV01C vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SCTV01C (Experimental)
  Interventions: Biological: SCTV01C
- SCTV01E (Experimental)
  Interventions: Biological: SCTV01E
- mRNA vaccine manufactured by Pfizer or Moderna (Active Comparator)
  Interventions: Biological: mRNA vaccine manufactured by Pfizer or Moderna
- Sinopharm inactivated COVID-19 vaccine (Active Comparator)
  Interventions: Biological: Sinopharm inactivated COVID-19 vaccine

INTERVENTIONS:
Biological: SCTV01C — Day 0; intramuscular injection
  Arms: SCTV01C
Biological: SCTV01C — Day 28; intramuscular injection
  Arms: SCTV01C
Biological: SCTV01C — Day 180; intramuscular injection
  Arms: SCTV01C
Biological: SCTV01E — Day 0; intramuscular injection
  Arms: SCTV01E
Biological: SCTV01E — Day 28; intramuscular injection
  Arms: SCTV01E
Biological: SCTV01E — Day 180; intramuscular injection
  Arms: SCTV01E
Biological: mRNA vaccine manufactured by Pfizer or Moderna — Day 0; intramuscular injection
  Arms: mRNA vaccine manufactured by Pfizer or Moderna
Biological: mRNA vaccine manufactured by Pfizer or Moderna — Day 28; intramuscular injection
  Arms: mRNA vaccine manufactured by Pfizer or Moderna
Biological: mRNA vaccine manufactured by Pfizer or Moderna — Day 180; intramuscular injection
  Arms: mRNA vaccine manufactured by Pfizer or Moderna
Biological: Sinopharm inactivated COVID-19 vaccine — Day 0; intramuscular injection
  Arms: Sinopharm inactivated COVID-19 vaccine
Biological: Sinopharm inactivated COVID-19 vaccine — Day 28; intramuscular injection
  Arms: Sinopharm inactivated COVID-19 vaccine
Biological: Sinopharm inactivated COVID-19 vaccine — Day 180; intramuscular injection
  Arms: Sinopharm inactivated COVID-19 vaccine

SUMMARY:
The objective of the study is to evaluate the immunogenicity and safety of SCTV01C or SCTV01E, comparing the immunogenicity data against Beta (B.1.351), Delta (B.1.617.2), Omicron (B.1.1.529) and other variants with Sinopharm inactivated COVID-19 vaccine or mRNA vaccine.

DETAILED DESCRIPTION:
The study is a randomized, double-blinded, active-controlled (Approved vaccine) Phase II clinical study. The study consists of 2 stages, Stage 1 and 2. In Stage 1, participants would randomly receive 2 doses of SCTV01C, SCTV01E, Sinopharm COVID-19 vaccine or mRNA vaccine on Day 0 and Day 28. Stage 1 is aimed to evaluate the immunogenicity and safety of SCTV01C or SCTV01E, comparing the immunogenicity data against Beta (B.1.351), Delta (B.1.617.2), Omicron (B.1.1.529) and other variants after the 2nd dose of vaccination with Sinopharm inactivated COVID-19 vaccine or mRNA vaccine. Stage 2 will start on Day 180 and the participants will receive a 3rd dose of vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥12 years old when signing ICF;
2. Participants who were neither vaccinated with any COVID-19 vaccine (including COVID-19 vaccine or vaccine adjuvant in clinical trial) nor diagnosed with COVID-19;
3. Participants or his/her legal guardian (or entrusted person) can sign written ICF and voluntarily participate in the trial, and can fully understand the trial procedure, the risk of participating in the trial, and other interventions that can be selected if they do not participate in the trial;
4. Participant him/herself or with the assistance of his/her family member is capable of finishing the record cards;
5. Healthy participants or participants with pre-existing medical conditions who are in stable condition. The "pre-existing medical conditions" include but not limited to hypertension, diabetes, chronic cholecystitis and cholelithiasis, chronic gastritis that meet the described criteria. A stable medical condition is defined as disease not requiring significant change in therapy or no need for hospitalization as a consequence of worsening disease state for at least 3 months prior to enrollment;
6. Fertile men and women of childbearing age voluntarily agree to take effective contraceptive measures from signing ICF to 6 months after the last dose of study vaccination; the pregnancy test results of women of childbearing age are negative on screening.

Exclusion Criteria:

1. Presence of fever within 3 days before the study vaccination;
2. A positive result of IgG antibody against the SARS-CoV-2 virus during the screen period;
3. A history of infection or disease related to severe acute respiratory syndrome (SARS), Middle East respiratory syndrome (MERS), or corresponding immunosuppressants;
4. A history of allergic reactions to any vaccine or drug, such as allergy, urticaria, severe skin eczema, dyspnea, laryngeal edema, and angioneurotic edema;
5. A medical or family history of seizure, epilepsy, encephalopathy and psychosis;
6. Immunocompromised patients suffering from immunodeficiency diseases, important organ diseases, immune diseases (including Guillain-Barre Syndrome [GBS], systemic lupus erythematosus, rheumatoid arthritis, asplenia or splenectomy caused by any circumstances, and other immune diseases that may have an impact on immune response in the investigator's opinion), etc.;
7. Long-term use of immunosuppressant therapy or immunomodulatory drugs for ≥14 days within the 1st six months prior to enrollment. Whereas short-term (≤14 days) use of oral, inhaled and topical steroids are allowed.
8. Patients on antituberculosis therapy;
9. Presence of severe or uncontrollable cardiovascular diseases, or severe or uncontrollable disorders related to endocrine system, blood and lymphatic system, liver and kidney, respiratory system, metabolic and skeletal systems, or malignancies (exception for skin basal cell carcinoma and carcinoma in-situ of cervix) , such as severe heart failure, severe pulmonary heart disease, unstable angina, liver failure, or uremia;
10. Contraindications for intramuscular injection or intravenous blood sampling, including thrombocytopenia and other blood coagulation disorders;
11. Participants who received any immunoglobulin or blood products in the previous 3 months, or plan to receive similar products during the study;
12. Participants who received other investigational drugs within 1 month before the study vaccination;
13. Participants who is at the acute state of disease, such as acute onset of chronic heart failure, acute sore throat, hypertensive encephalopathy, acute pneumonia, acute renal insufficiency, acute cholecystitis;
14. Participants received other drugs used for prevention of COVID-19;
15. Participants vaccinated with influenza vaccine within 14 days or with other vaccines within 28 days before the study vaccination;
16. Those who donated blood or had blood loss (≥450 mL) within 3 months before the vaccination or plan to donate blood during the study period;
17. Those who are pregnant or breast-feeding or plan to be pregnant during the study period;
18. Those who plan to donate ovum or sperms during the study period;
19. Those who cannot follow the trial procedures, or cannot cooperate to complete the study due to planned relocation or long-term outing;
20. Those unsuitable for participating in the clinical trial as determined by the investigator because of other abnormalities that are likely to confuse the study results, or non-conformance with the maximal benefits of the participants;
21. Those who are tested positive for HIV in terms of serology.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Geometric mean titers (GMT) of neutralizing antibody against Beta (B.1.351) variant on Day 56 (28 days after the 2nd dose of vaccination); | Day 56 after the study vaccination
Stage 1: GMT of neutralizing antibody against Delta (B.1.617.2) variant on Day 56 (28 days after the 2nd dose of vaccination); | Day 56 after the study vaccination
Stage 1: GMT of neutralizing antibody against Omicron (B.1.1.529) variant on Day 56 (28 days after the 2nd dose of vaccination); | Day 56 after the study vaccination
Stage 2: GMT of neutralizing antibody against Beta (B.1.351) variant on Day 208 (28 days after the 3rd dose of vaccination); | Day 208 after the study vaccination
Stage 2: GMT of neutralizing antibody against Delta (B.1.617.2) variant on Day 208 (28 days after the 3rd dose of vaccination); | Day 208 after the study vaccination
Stage 2: GMT of neutralizing antibody against Omicron (B.1.1.529) variant on Day 208 (28 days after the 3rd dose of vaccination); | Day 208 after the study vaccination
Incidence and severity of solicited AEs within 7 days after each dose of vaccine (Day 0 to Day 7, Day 28 to Day 35, and Day 180 to Day 187). | 7 days after each study vaccination

SECONDARY OUTCOMES:
Stage 1: GMT of neutralizing antibody against Beta (B.1.351) variant on Day 180 (before the injection of the 3rd dose of vaccination); | Day 180 after the study vaccination
Stage 1: GMT of neutralizing antibody against Delta (B.1.617.2) variant on Day 180 (before the injection of the 3rd dose of vaccination); | Day 180 after the study vaccination
Stage 1: GMT of neutralizing antibody against Omicron (B.1.1.529) variant on Day 180 (before the injection of the 3rd dose of vaccination); | Day 180 after the study vaccination
Stage 1: Number of IFN-γ positive (characterizing Th1) and IL-4 positive (characterizing Th2) T cell subpopulations on Day 0, Day14, Day 28 and Day 42; | Day 0, Day 14, Day 28 and Day 42 after the study vaccination
Stage 1: Seroresponse rates of neutralizing antibodies to Beta [B.1.351], Delta [B.1.617.2] and Omicron [B.1.1.529] variants on Day 56; | Day 56 after the study vaccination
Stage 2: GMT of neutralizing antibody against Beta (B.1.351) variant on Day 365 (185 days after the 3rd dose of vaccination); | Day 365 after the study vaccination
Stage 2: GMT of neutralizing antibody against Delta (B.1.617.2) variant on Day 365 (185 days after the 3rd dose of vaccination); | Day 365 after the study vaccination
Stage 2: GMT of neutralizing antibody against Omicron (B.1.1.529) variant on Day 365 (185 days after the 3rd dose of vaccination); | Day 365 after the study vaccination
Stage 2: Number of IFN-γ positive (characterizing Th1) and IL-4 positive (characterizing Th2) T cell subpopulations on Day 180 (Before the injection of the 3rd dose of vaccination) and Day 194 (14 days after the 3rd dose of vaccination); | Day 180 (Before the injection of the 3rd dose of vaccination) and Day 194 (14 days after the 3rd dose of vaccination)
Stage 2: Seroresponse rates of neutralizing antibodies to Beta [B.1.351], Delta [B.1.617.2] and Omicron [B.1.1.529] variants on Day 208; | Day 208 after the study vaccination
Incidence and severity of unsolicited systemic AEs within 28 days after each dose of vaccine (Day 0 to Day 28, Day 28 to Day 56, and Day 180 to Day 208); | 28 days after each study vaccination
Incidence and severity of serious adverse events (SAEs) and adverse events of special interest (AESIs) within 365 days after the 1st dose of vaccination. | Day 0 to Day 365 after the study vaccination